CLINICAL TRIAL: NCT01020370
Title: An Exploratory Study to Investigate the Reparative and Regenerative Potential of Alemtuzumab in Relapsing-Remitting Multiple Sclerosis: A Multi-Parametric Non-Conventional MRI Sub-Study in Patient Participating in the CARE MS I and CARE MS II Studies
Brief Title: Exploratory Study to Investigate the Reparative and Regenerative Potential of Alemtuzumab in Relapsing-Remitting Multiple Sclerosis Patients Participating in the CARE MS I and MS II Studies
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Other Study IDs: CAMMS030081ST
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Multiple Sclerosis
Keywords: Patients with RRMS who are participating in the CARE MS I and CARE MS II
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Alemtuzumab Group
- Interferon Beta-1a SC Group

SUMMARY:
The primary goal of this study will be to explore the reparative and regenerative potential of alemtuzumab in RRMS patients who are participating in the CARE MS I and CARE MS II studies using conventional and non-conventional MRI sequences.

ELIGIBILITY:
Inclusion Criteria:

* Participating in either the CARE MS I or CARE MS II studies

Exclusion Criteria:

* Not a participant in the CARE MS I or CARE MS II studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RRMS who are participating in the CARE MS I and CARE MS II studies and are receiving either alemtuzumab or interferon beta-1a SC
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Explore the reparative and regenerative potential of alemtuzumab in RRMS patients who are participating in the CARE MS I and CARE MS II studies

SECONDARY OUTCOMES:
Compare the effect of alemtuzumab to interferon beta-1a SC on non-conventional MRI outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Omar Khan, MD, Principal Investigator — Wayne State University